CLINICAL TRIAL: NCT05005637
Title: Antitubercular Treatment for Uveitis of Undetermined Cause with Positive QuantiFERON-TB Gold Plus: a Randomized Clinical Trial
Brief Title: The Effectivity of Anti Tuberculosis Therapy in Idiopathic Uveitis with Positive IGRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Rina, Staff of Ocular Infection and Immunology Department, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06/DIPI/2021
Record Dates: First submitted 2021-08-10; First posted 2021-08-13 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Tuberculous Uveitis
Keywords: Tuberculosis; Uveitis; Tuberculous Uveitis; Idiopathic Uveitis; Interferon Gamma Release Assay; Anti Tuberculosis Therapy; IGRA; ATT; Quantiferon-TB GoldPlus
MeSH Terms: conditions — Tuberculosis; Uveitis | interventions — Antitubercular Agents; Methylprednisolone

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti Tuberculosis Therapy (Experimental): Dosage form: ATT fixed-dose combination (FDC). FDC intensive phase containing 150 mg of rifampicin, 75 mg of isoniazid not 300mg, 400 mg of pyrazinamide, and 275 mg of ethambutol, while FDC continuation phase containing rifampicin-isoniazid.
  Dosage: according to body weight, 30-37 kg: 2 tablets, 38-54 kg: 3 tablets, 55-70 kg: 4 tablets, more than 70 kg: 5 tablets.
  Frequency: Intensive phase: once daily. Continuation phase: 3 times/week. Duration: 9 months (2 months of FDC intensive phase + 7 months of FDC continuation phase)
  Interventions: Drug: Anti Tuberculosis Drug
- Steroid Local and Oral (Active Comparator): Local steroids were prescribed according to the standard care by the attending uveitis specialists and tailored to the severity of the intraocular inflammation. Additionally, all participants in this group received oral methylprednisolone at a dosage of 0.8 mg/kg of body weight per day (maximum of 56 mg/day), which was tapered gradually based on the intraocular inflammation observed. Tapering of oral methylprednisolone involved reducing the dose by 8 mg for doses above 20 mg and by 4 mg for doses below 20 mg.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Anti Tuberculosis Drug — ATT will be given in the form of fixed drug combination (FDC). Each patient will get a regimen of 2RHZE (2 months of FDC intensive phase, which contains of Rifampicin, Isoniazide, Pirazinamide, Ethambutol) + 7RH (7 months of FDC continuation phase, which contains of Rifampicin and Isoniazid). The dosage will be according to body weight, 30-37 kg: 2 tablets, 38-54 kg: 3 tablets, 55-70 kg: 4 tablets, more than 70 kg: 5 tablets. FDC drugs have to be consumed daily during intensive phase and three times a week during continuation phase.
  Arms: Anti Tuberculosis Therapy
Drug: Methylprednisolone — Selected participants may be prescribed local or systemic immunosuppressants, including oral methylprednisolone, starting at a dosage of 0.8 mg/kg of body weight per day and tapered gradually (e.g., every three days or weekly) based on the severity of intraocular inflammation observed during presentation and follow-up visits.
  Arms: Steroid Local and Oral

SUMMARY:
The reported incidence of uveitis is 52 persons per year per 100,000 population, with a greater incidence estimated in developing countries, including Indonesia. Uveitis has challenges in diagnosis and therapy, due to the existence of an immunological privilege mechanism, so it is not easy to obtain diagnostic markers or provide appropriate therapy. In uveitis, a work-up examination looking for signs in the entire body or systemic disease is often conducted.

Up until today, establishing the diagnosis of tuberculosis (TB)-associated uveitis is still a challenge. From histopathological studies, TB germs are difficult to find. Wreblowski et al. found that paucibacillary conditions also made TB bacteria difficult to find by PCR and tuberculin test results were also not completely reliable. The development of IGRA (Interferon-Gamma Release Assay) assays, such as QuantiFERON-Gold TB (QFT) has been investigated. Our previous study found that IGRA-positive uveitis patients with type 1 IFN gene expression score >5.61 were more likely to have active TB uveitis. In addition, serum C1q examination also showed an inverse correlation with this score.

Regarding therapy, until now corticosteroids and cycloplegics are the mainstay treatment for uveitis. However, appropriate administration of anti-infective drugs is necessary in cases of infection. Inflammation in TB-associated uveitis is thought to be the result of the immune response that occurs as a result of paucibacillary TB infection. Examinations can be redundant and problematic. Determination of therapy is also a dilemma because it is difficult to determine the right patient candidate for administration of anti-tuberculosis therapy (ATT). The protocol of ATT administration itself has not been standardized so it often follows the extra pulmonary TB protocol and there has been no reliable clinical trial research on ATT administration in patients with suspected TB uveitis yet no TB microorganisms are found directly in the eyes or other organs.

On this basis, the investigators planned a prospective randomized clinical trial study that involve idiopathic uveitis patients with positive IGRA test, to assess the effectivity of ATT compared to oral steroids. In addition, this study can also be used as a basis for validation of type 1 IFN scores and serum C1q as diagnostic/prognostic biomarkers in cases of TB-associated uveitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient that is newly diagnosed with uveitis of unknown origin/idiopathic (as evidenced by a series of uveitis work-up tests) and tested positive for IGRA (>0.35 U/ml).
2. Age >18 years old
3. Lives in Jakarta/Bogor/Depok/Tangerang/Bekasi area or willing to participate in research until the end of monitoring program
4. Willing to participate in the research and sign the informed consent after receiving explanation regarding the research

Exclusion Criteria:

1. Patients with positive aqueous tap examination results on one of the examination panels for the bacteria causing infectious uveitis according to the standard examination
2. Anterior uveitis patient with a positive HLA-B27 test result
3. The patient is proven to have active TB or lives in the same house with an active TB patient
4. Patients are included in the TB reactivation risk index group according to the 2018 WHO LTBI (Latent Tuberculosis Incident) Guideline
5. HIV positive patient
6. Patients with uveitis sanata at the first visit
7. Patients with visual acuity less than 1/300 or showing signs of preptisis based on ophthalmological examination and ultrasound of the eye
8. The patient has a history of previous ATT consumption
9. Patients with impaired liver function or other systemic conditions which according to the Internal Medicine Department are not eligible to receive ATT
10. The patient has a history of taking antibiotics in the last 1-2 weeks
11. The patient is not willing to sign the informed consent
12. The patient was pregnant at the first visit or was planning to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Treatment Failure | 6 months after the initial therapy
  Treatment will be categorized as a failure if subject did not meet the following criteria at the 6-month follow-up post initial therapy, (1) less than or equal to 0.5+ anterior chamber cells by SUN criteria, less than or equal to 0.5+ vitreous haze clinical grading using the NEI scale, and no active retinal or choroidal lesions; and (2) no more than 7.5 mg of oral prednisone daily and less than or equal to 2 drops of prednisolone acetate 1% (or equivalent) per day; or in other words, the subject has persistent inflammation that keeps getting worse.
Response to Treatment | 6 months after initial treatment
  Criteria for complete uveitis resolution applied to both eyes, in cases with bilateral uveitis, included: (1) fewer than or equal to 0.5+ anterior chamber cells according to the Standardized Uveitis Nomenclature (SUN) grading system, fewer than or equal to 0.5+ vitreous haze based on clinical grading using the NEI (National Eye Institute) scale, and no active retinal or choroidal lesions; and (2) no more than 7.5 mg of oral prednisone daily (i.e., methylprednisolone at 6 mg or less daily) and fewer than or equal to 2 drops of prednisolone acetate 1% (or equivalent) per day. Treatment will be categorized as a failure if subject did not meet the following criteria at the 6-month follow-up.

SECONDARY OUTCOMES:
Time to Uveitis Resolution | 90 days after the visit of first uveitis resolution was recorded
  Calculated from the time of randomization. These criteria had to be maintained for at least 90 days following the visit when the first complete uveitis resolution was recorded. If there was insufficient follow-up after resolution, maintained uveitis resolution was still considered. Participants who met criterion 1 but not criterion 2 were classified as having partial uveitis resolution (non-complete uveitis resolution).
  This was measured every visit using objectives of ophthalmologist's clinical judgement from slit-lamp examination and clinical complaints.
Uveitis Relapse | 6 months after the initial therapy
  Uveitis relapse was defined as any worsening of ocular inflammation (including a two-step increase in anterior chamber or vitreous cells as per the SUN grading system) or the occurrence of clinically new inflammatory activity (such as choroidal or retinal lesions) that necessitated a modification of local or systemic uveitis treatment after a minimum of 90 days of complete uveitis resolution at the patient level.
  Time to relapse was calculated from the first visit showing inactive uveitis until the first notification of uveitis relapse.
Eye-Level outcome (Visual Acuity) | 6 months after baseline visit
  The differences in visual acuity between baseline and month 6.Visual acuity was considered to increase if the difference in best-corrected visual acuity between month 6 and baseline visits (measured with Snellen, in decimal equivalent) was equal to or greater than 0.1, stable if within the range of -0.1 to 0.1, and decreased if less than -0.1. If any cataract or vitreoretinal surgery was performed before the six-month follow-up, the last recorded visual acuity prior to the surgery was used.
Eye-Level outcome (Secondary glaucoma) | 6 months after baseline visit
  The incidence of secondary glaucoma (e.g., occurrences of increased intraocular pressure (IOP) above 21 mmHg in at least two consecutive visits that necessitated prescription of IOP-lowering medications).

CONTACTS AND LOCATIONS:
Overall Officials: Rina La Distia Nora, MD, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo National Central General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Putera I, Ten Berge JCEM, Thiadens AAHJ, Dik WA, Agrawal R, van Hagen PM, La Distia Nora R, Rombach SM. Relapse in ocular tuberculosis: relapse rate, risk factors and clinical management in a non-endemic country. Br J Ophthalmol. 2024 Nov 22;108(12):1642-1651. doi: 10.1136/bjo-2024-325207. PMID 38609164
- [Background] Putera I, Ten Berge JCEM, Thiadens AAHJ, Dik WA, Agrawal R, van Hagen PM, La Distia Nora R, Rombach SM. Clinical Features and Predictors of Treatment Outcome in Patients with Ocular Tuberculosis from the Netherlands and Indonesia: The OculaR TB in Low versus High Endemic Countries (ORTEC) Study. Ocul Immunol Inflamm. 2025 Jan;33(1):86-97. doi: 10.1080/09273948.2024.2359614. Epub 2024 May 31. PMID 38820475
- [Background] Putera I, Schrijver B, Ten Berge JCEM, Gupta V, La Distia Nora R, Agrawal R, van Hagen PM, Rombach SM, Dik WA. The immune response in tubercular uveitis and its implications for treatment: From anti-tubercular treatment to host-directed therapies. Prog Retin Eye Res. 2023 Jul;95:101189. doi: 10.1016/j.preteyeres.2023.101189. Epub 2023 May 25. PMID 37236420
- [Background] Ludi Z, Sule AA, Samy RP, Putera I, Schrijver B, Hutchinson PE, Gunaratne J, Verma I, Singhal A, Nora RD, van Hagen PM, Dik WA, Gupta V, Agrawal R. Diagnosis and biomarkers for ocular tuberculosis: From the present into the future. Theranostics. 2023 Apr 1;13(7):2088-2113. doi: 10.7150/thno.81488. eCollection 2023. PMID 37153734
- [Background] La Distia Nora R, Sitompul R, Bakker M, Susiyanti M, Edwar L, Sjamsoe S, Singh G, van Hagen MP, Rothova A. Tuberculosis and other causes of uveitis in Indonesia. Eye (Lond). 2018 Mar;32(3):546-554. doi: 10.1038/eye.2017.231. Epub 2017 Nov 3. PMID 29099497
- [Background] Betzler BK, Putera I, Testi I, La Distia Nora R, Kempen J, Kon OM, Pavesio C, Gupta V, Agrawal R. Anti-tubercular therapy in the treatment of tubercular uveitis: A systematic review and meta-analysis. Surv Ophthalmol. 2023 Mar-Apr;68(2):241-256. doi: 10.1016/j.survophthal.2022.10.001. Epub 2022 Oct 19. PMID 36272559
- [Derived] La Distia Nora R, Putera I, Riasanti M, Sitompul R, Edwar L, Susiyanti M, Aziza Y, Waliyuddin MZ, Widodo E, Sifyana UA, Jessica P, Ethelind R, Singh G, Dik WA, Rombach SM, van Hagen PM. Antitubercular therapy for uveitis of undetermined cause with positive interferon-gamma release assay: a single-blind, single-centre, phase 2 randomised controlled trial. EClinicalMedicine. 2025 Sep 17;88:103511. doi: 10.1016/j.eclinm.2025.103511. eCollection 2025 Oct. PMID 41018498